CLINICAL TRIAL: NCT07402213
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of JYB1904 Injection in Adult Patients With Chronic Spontaneous Urticaria Inadequately Controlled by H1 Antihistamines
Brief Title: Trial of JYB1904 Injection in Adult Patients With Chronic Spontaneous Urticaria.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JYB1904-301
Record Dates: First submitted 2026-01-28; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: CSU
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JYB1904 Injection Group (Experimental): 300 mg JYB1904 injection administered SC
  Interventions: Drug: JYB1904
- Placebo Group (Placebo Comparator): Placebo and 300 mg JYB1904 injection administered SC
  Interventions: Drug: Placebo+JYB1904

INTERVENTIONS:
Drug: JYB1904 — 300 mg JYB1904 injection administered SC every 12 weeks (Q12W) from Day 1 to Week 48.
  Other Names: JYB1904 Injection
  Arms: JYB1904 Injection Group
Drug: Placebo+JYB1904 — Placebo administered SC on D1 and W12; 300 mg JYB1904 injection administered SC every 12 weeks (Q12W) from W24 to W48.
  Other Names: Placebo+JYB1904 Injection
  Arms: Placebo Group

SUMMARY:
This Phase III Trial is Meant to Evaluate the Efficacy, and Safety of JYB1904 Injection in Adult Patients With Chronic Spontaneous Urticaria.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, placebo-controlled Phase III study to evaluate the efficacy and safety of JYB1904 injection compared to placebo in patients with CSU inadequately controlled by second-generation H1 antihistamines.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant must be ≥18 years old at the time of signing the informed consent.
* Participants are diagnosed with CSU for ≥6 months before screening.
* Participants suffer from itching and hives for at least 6 consecutive weeks at any time before screening.
* UAS7 (range 0~42) ≥16, ISS7 (range 0~21) ≥8 during 7 days before randomization.
* Participants treated with stable dose of second-generation H1 antihistamines (up to 4x approved dose) for at least 6 consecutive weeks before randomization, switching medications, or changing drug dosage or frequency is not allowed within 3 weeks before randomization.
* Participants have ≥6 days record of UAS7 before randomization.

Exclusion Criteria:

* Participants who suffer from inducible urticaria with definite inducements, including urticaria factitia (dermatographism), cold contact, heat contact, solar, pressure, delayed pressure, aquagenic, cholinergic or contact urticaria, etc.
* Participants who suffer from any other skin diseases with chronic itching, such as atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus or psoriasis, etc.
* Participants who suffer from other diseases with symptoms of urticaria or angioedema, including but not limited to urticaria vasculitis, urticaria pigmentosa, erythema multiforme, mastocytosis, hereditary urticaria or acquired/drug-induced urticaria.
* Participants who are contraindicated or hypersensitive to antihistamines or any of its component (such as fexofenadine, loratadine, desloratadine, cetirizine, levocetirizine, rupatadine, bilastine).
* History of anaphylactic shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-04-28 (Estimated)

PRIMARY OUTCOMES:
Urticaria Activity Score Over 7 Consecutive Days(UAS7) | Up to 12 weeks
  Change from baseline in UAS7 at W12.
  The UAS7 is a composite score derived from the ISS7 and the HSS7, i.e., the sum of ISS7 and HSS7, ranging from 0 to 42 points. UAS7 = 0 indicates complete resolution of urticaria.

SECONDARY OUTCOMES:
Itch Severity Score Over 7 Consecutive Days(ISS7) | Up to 12 weeks
  Change from baseline in ISS7 at W12.
  The ISS7 is the sum of mean daily scores over the 7 days prior to the visit, ranging from 0 to 21 points. ISS7 = 0 indicates complete resolution of itch.
Urticaria Activity Score Over 7 Consecutive Days(UAS7) | Up to 12 weeks
  Proportion of participants with UAS7=0 at W12
Urticaria Activity Score Over 7 Consecutive Days(UAS7) | Up to 24 weeks
  Change from baseline in UAS7 at W24
Urticaria Activity Score Over 7 Consecutive Days(UAS7) | Up to 24 weeks
  Proportion of participants with UAS7=0 at W24
Itch Severity Score Over 7 Consecutive Days(ISS7) | Up to 24 weeks
  Change from baseline in ISS7 at W24
Hive Severity Score Over 7 Consecutive Days (HSS7) | Up to 24 weeks
  Change from baseline in HSS7 at W12 and W24.
  The HSS7 is the sum of mean daily scores over the 7 days prior to the visit, ranging from 0 to 21 points. HSS7 = 0 indicates complete resolution of hives.
Angioedema Activity Score Over 7 Consecutive Days(AAS7) | Up to 24 weeks
  Change from baseline in AAS7 at W12 and W24. The AAS7 is the sum of the daily scores over the 7 days prior to the visit, ranging from 0 to 105 points.AAS7 = 0 indicates no angioedema.
Urticaria Activity Score Over 7 Consecutive Days(UAS7) | Up to 24 weeks
  Proportion of participants with UAS7≤ 6 at W12 and W24
Dermatology Life Quality Index(DLQI) | Up to 24 weeks
  Change from baseline in DLQI at W12 and W24.
  The DLQI comprises 10 questions that assess the participant's skin symptoms and the impact of their dermatological condition on multiple life domains over the past 7 days. The total score ranges from 0 to 30. The higher the score, the worse the quality of life.
Efficacy Assessment Scale | Through study completion, an average of 72 weeks
  Change from baseline in UAS7, ISS7, HSS7, AAS7 (AAS7 only in participants with baseline AAS7>0) over time during the study
Efficacy Assessment Scale | Through study completion, an average of 72 weeks
  Proportion of participants with UAS7=0, ISS7=0, HSS7=0, AAS7=0 (AAS7 only in participants with baseline AAS7>0) over time during the study
Urticaria Activity Score Over 7 Consecutive Days(UAS7) | Through study completion, an average of 72 weeks
  Proportion of participants with UAS7≤ 6 over time during the study
Dermatology Life Quality Index(DLQI) | Through study completion, an average of 72 weeks
  Change from baseline in DLQI over time during the study
Dermatology Life Quality Index(DLQI) | Through study completion, an average of 72 weeks
  Proportion of participants with DLQI=0/1 over time during the study
Urticaria Activity Score Over 7 Consecutive Days(UAS7) | Up to 24 weeks
  Cumulative number of weeks with UAS7 ≤ 6 by W12 and W24
Angioedema Activity Score Over 7 Consecutive Days(AAS7) | Up to 24 weeks
  Cumulative number of weeks with AAS7 = 0 by W12 and W24
Rescue Therapy | Up to 24 weeks
  Proportion of participants requiring rescue therapy by W12 and W24
Safety and tolerability | Through study completion, an average of 72 weeks
  Adverse events (AEs) and serious adverse events (SAEs), vital signs, physical examination, 12-lead electrocardiogram (ECG) and laboratory results

OTHER OUTCOMES:
Pharmacokinetic (PK) profile of JYB1904 injection | Through study completion, an average of 72 weeks
  Serum concentration of JYB1904
Pharmacodynamic (PD) profile of JYB1904 injection | Through study completion, an average of 72 weeks
  PD parameters: Changes in serum level of total and free IgE
Immunogenicity of JYB1904 injection | Through study completion, an average of 72 weeks
  Immunogenicity parameters: Positive detection rate of anti-drug antibodies (ADA)/neutralizing ADA (Nab), ADA onset time, duration, and titer

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, Principal Investigator — Peking University People's Hospital; Cheng Zhou, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No